CLINICAL TRIAL: NCT00098787
Title: Phase II Study of Treatment Selection Based Upon Tumor Thymidylate Synthase Expression in Previously Untreated Patients With Metastatic Colorectal Cancer
Brief Title: Bevacizumab and Oxaliplatin Combined With Irinotecan or Leucovorin and Fluorouracil in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000398096; E4203 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (High TS, IROX/bev) (Experimental): Patients with high TS who are randomized to Arm A receive irinotecan and oxaliplatin plus bevacizumab (IROX/bev). The combination regimen is administered by giving bevacizumab IV over 30-90 minutes followed by oxaliplatin IV over 2 hours and irinotecan IV over 90 minutes on days 1 and 15 every 28 days until disease progression or until any criterion specified in protocol is met.
  Interventions: Biological: bevacizumab; Drug: irinotecan hydrochloride; Drug: Oxaliplatin
- Arm B (High TS, FOLFOX/bev) (Experimental): Patients with high TS who are randomized to Arm B receive 5-Fluorouracil, leucovorin, oxaliplatin, and bevacizumab (FOLFOX/bev). The combination regimen is administered by giving bevacizumab and oxaliplatin as in Arm A, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15 every 28 days until disease progression or until any criterion specified in protocol is met.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: Oxaliplatin
- Arm C (Low or intermediate TS, FOLFOX/bev) (Experimental): Patients with low or intermediate TS receive 5-Fluorouracil, leucovorin, oxaliplatin, and bevacizumab (FOLFOX/bev) as in Arm B.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: Oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: NSC 704865, RhuMAb VEGF, Recombinant Humanized Monoclonal Anti-VEGF Antibody
Drug: fluorouracil — Given IV
  Other Names: 5-Fluorouracil, 5-FU, Adrucil, Efudex
  Arms: Arm B (High TS, FOLFOX/bev); Arm C (Low or intermediate TS, FOLFOX/bev)
Drug: irinotecan hydrochloride — Given IV
  Other Names: Camptothecin-11, CPT-11, Camptosar
  Arms: Arm A (High TS, IROX/bev)
Drug: leucovorin calcium — Given IV
  Other Names: Leucovorin, Wellcovorin' citrovorum factor, folinic acid, 5-formyl tetrahydrofolate, LV, LCV.
  Arms: Arm B (High TS, FOLFOX/bev); Arm C (Low or intermediate TS, FOLFOX/bev)
Drug: Oxaliplatin — Given IV
  Other Names: Eloxatin, trans-l-diaminocyclohexane oxalatoplatinum, cis-[oxalato(trans-l-1,2-diaminocyclohexane)platinum(II)].

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, irinotecan, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. Giving bevacizumab together with combination chemotherapy may be a better way to block tumor growth. Studying the amount of an enzyme found in the tumor may help doctors plan the best treatment.

PURPOSE: This randomized phase II trial is studying giving bevacizumab, oxaliplatin, and irinotecan or giving bevacizumab, oxaliplatin, leucovorin, and fluorouracil in treating patients with metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate (complete and partial), progression-free survival, and overall survival of patients with previously untreated metastatic or locally recurrent colorectal adenocarcinoma with high vs low thymidylate synthase (TS) expression treated with fluorouracil, leucovorin calcium, oxaliplatin, and bevacizumab or irinotecan, oxaliplatin, and bevacizumab.
* Compare the toxicity of these regimens in these patients.
* Correlate gene expression with response rates in patients treated with these regimens.
* Correlate gene expression with toxicity of these regimens in these patients.
* Correlate dihydropyrimidine dehydrogenase, thymidine phosphorylase, and mammalian excision repair cross complementary protein expression with antitumor response in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to thymidylate synthase (TS) expression levels (high vs low or indeterminate). Patients with high TS expression are randomized to 1 of 2 treatment arms (Arms A or B). Patients with low or indeterminate TS expression are assigned to Arm C.

* Arm A: Patients receive bevacizumab IV over 30-90 minutes followed by oxaliplatin IV over 2 hours and irinotecan IV over 90 minutes on days 1 and 15.
* Arm B: Patients receive bevacizumab and oxaliplatin as in arm A, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15.
* Arm C: Patients receive bevacizumab, oxaliplatin, leucovorin calcium, and fluorouracil as in arm B.

In all arms, courses repeat every 28 days in the absence of unacceptable toxicity or disease progression.

Patients are followed up every 3 months for 2 years and then every 6 months for 2 years from the date of study registration.

ELIGIBILITY:
INCLUSION:

* Metastatic or locally recurrent colorectal adenocarcinoma
* Measurable disease
* At least 2 formalin-fixed paraffin embedded core needle biopsies OR fine needle aspirate containing a minimum of 3 clusters of malignant cells and fixed tissue from the previous biopsy
* If no tissue samples are available the patient must be willing to undergo biopsy of a metastatic site
* Age 18 and over
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Prothrombin time (PT)/international normalized ratio (INR) ≤ 1.5 unless patient is receiving full-dose anticoagulants AND the following criteria are met:

  * In-range INR (usually between 2 and 3) AND on a stable dose of warfarin or low molecular weight heparin
  * No active bleeding or pathological condition that is associated with a high risk of bleeding
* Partial thromboplastin time (PTT) < 1.5 times upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) < 3 times ULN
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.8 mg/dL
* Meets 1 of the following criteria:

  * Protein negative on urine dipstick
  * Urine protein/creatinine ratio < 1.0
  * Less than 2 g protein on 24-hour urine collection
* Patients with a history of hypertension must meet the following criteria:

  * Blood pressure < 150/90 mm Hg
  * Stable regimen of anti-hypertensive therapy
* More than 28 days since prior major or open surgery
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* Prior non-colorectal malignancies are allowed provided the following criteria are met:

  * No current clinical evidence of persistent or recurrent disease
  * No active therapy for non-colorectal malignancy, including hormonal therapy

EXCLUSION:

* Pregnant or nursing
* Arterial thromboembolic events within the past 6 months, including the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina pectoris
  * Myocardial infarction
* Symptomatic arrhythmia
* Symptomatic congestive heart failure
* Clinically significant peripheral artery disease
* New York Heart Association class III or IV heart disease
* Serious nonhealing wound, ulcer, or bone fracture within the past 28 days
* Significant traumatic injury within the past 28 days
* Neuropathy ≥ grade 2
* Ongoing or active infection
* Concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* Prior chemotherapy for metastatic disease. Adjuvant therapy completed at least 12 months before first evidence of metastasis allowed
* Cardiovascular, renal, hepatic, or other nonmalignant systemic disease that would preclude study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2005-09-08 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Study Chair — Fox Chase Cancer Center; Jean L. Grem, MD, Study Chair — University of Nebraska
Locations (110):
- United States (110):
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on July 14, 2005, accrued its first patient on September 8, 2005, and terminated on April 20, 2012, with 247 patients from 25 institutions enrolled to the study.
Pre-assignment Details: Only 211 patients were registered to the treatment phase of the study, while the other 36 did not proceed because of ineligibility (n=9), patient withdrawal (n=6), unknown thymidylate synthase (TS)/insufficient sample (n=3), disease progression/decline in TS (n=2), Arm C suspended could not enter Step 2 (n =15), and no insurance (n =1).
Period: Overall Study
Arm/Group | Arm A (High TS, IROX/Bev) | Arm B (High TS, FOLFOX/Bev) | Arm C (Low or Intermediate TS, FOLFOX/Bev)
Started | 73 | 75 | 63
Treated | 70 | 73 | 62
Eligible and Treated | 61 | 66 | 59
Completed | 0 | 0 | 0
Not Completed | 73 | 75 | 63
Not completed — Never started treatment | 3 | 2 | 1
Not completed — Ineligible | 9 | 7 | 3
Not completed — Disease progression | 28 | 17 | 23
Not completed — Adverse Event | 8 | 17 | 8
Not completed — Death | 6 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 12 | 6
Not completed — Alternative therapy | 8 | 13 | 13
Not completed — Other | 7 | 6 | 9

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (High TS, IROX/Bev) | Arm B (High TS, FOLFOX/Bev) | Arm C (Low or Intermediate TS, FOLFOX/Bev) | Total
Number analyzed (Participants) | 61 | 66 | 59 | 186
Age, Continuous [Median (Full Range); unit: years] | 61 [37 to 85] | 60 [31 to 79] | 59 [29 to 80] | 60 [29 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 30 | 24 | 75
  Male | 40 | 36 | 35 | 111
Disease status [Number; unit: participants]
  Initial Diagnosis | 50 | 50 | 50 | 150
  Recurrence | 11 | 16 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is defined as proportion of patients who achieve complete response (CR) or partial response (PR). Response was assessed using Solid Tumor Response Criteria (RECIST). CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Assessed every 3 months if the patient is within 2 years of registration and every 6 months up to 4 years post-registration.
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: proportion
Arm/Group | Arm A (High TS, IROX/Bev) | Arm B (High TS, FOLFOX/Bev) | Arm C (Low or Intermediate TS, FOLFOX/Bev)
Number analyzed (Participants) | 61 | 66 | 59
proportion | 0.33 [0.23 to 0.44] | 0.38 [0.28 to 0.49] | 0.49 [0.38 to 0.61]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival is defined as time from randomization (to Arm A or Arm B) or registration (to Arm C) to the earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored.
Time Frame: Assessed every 3 months if the patient is within 2 years of registration and every 6 months once the patient is 2-4 years post-registration.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (High TS, IROX/Bev) | Arm B (High TS, FOLFOX/Bev) | Arm C (Low or Intermediate TS, FOLFOX/Bev)
Number analyzed (Participants) | 61 | 66 | 59
months | 10 [6 to 11] | 9 [8 to 11] | 13 [10 to 14]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from randomization (to Arm A or Arm B) or registration (to Arm C) to death. Patients alive at last follow-up were censored.
Time Frame: as for outcome 2
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (High TS, IROX/Bev) | Arm B (High TS, FOLFOX/Bev) | Arm C (Low or Intermediate TS, FOLFOX/Bev)
Number analyzed (Participants) | 61 | 66 | 59
months | 18 [14 to 23] | 21 [16 to 32] | 32 [23 to 44]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment
Groups:
- High TS: IROX/Bev: Patients with high thymidylate synthase (TS) who are randomized to Arm A receive irinotecan and oxaliplatin plus bevacizumab (IROX/bev). The combination regimen is administered by giving bevacizumab IV over 30-90 minutes followed by oxaliplatin IV over 2 hours and irinotecan IV over 90 minutes on days 1 and 15 every 28 days until disease progression or until any criterion specified in protocol.
- High TS: FOLFOX/Bev: Patients with high thymidylate synthase (TS) who are randomized to Arm B receive 5-Fluorouracil, leucovorin, oxaliplatin, and bevacizumab (FOLFOX/bev). The combination regimen is administered by giving bevacizumab and oxaliplatin as in arm I, leucovorin calcium IV over 2 hours, and fluorouracil IV over 5 minutes and then continuously over 46 hours on days 1 and 15 every 28 days until disease progression or until any criterion specified in protocol is met.
- Low or Indeterminate TS: FOLFOX/Bev: Patients with low or intermediate thymidylate synthase (TS) receive 5-Fluorouracil, leucovorin, oxaliplatin, and bevacizumab (FOLFOX/bev) as in Arm B.
Arm/Group | High TS: IROX/Bev | High TS: FOLFOX/Bev | Low or Indeterminate TS: FOLFOX/Bev
Serious Adverse Events (participants affected / at risk) | 49/70 | 53/73 | 43/62
Other Adverse Events (participants affected / at risk) | 70/70 | 73/73 | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High TS: IROX/Bev (N=70) | High TS: FOLFOX/Bev (N=73) | Low or Indeterminate TS: FOLFOX/Bev (N=62)
Anaphylaxis (Immune system disorders) | 2 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 2
White blood cell decreased (Investigations) | 12 | 4 | 7
Neutrophil count decreased (Investigations) | 16 | 28 | 21
Platelet count decreased (Investigations) | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 4 | 5
Hypotension (Vascular disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0
Fatigue (General disorders) | 15 | 7 | 4
Chills (General disorders) | 1 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Death NOS (General disorders) | 1 | 0 | 0
Sudden death NOS (General disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 9 | 2 | 7
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Colonic obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 3 | 2
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Infections and infestations - Other, spe (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, spe (Infections and infestations) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0
Infections and infestations - Other, spe (Infections and infestations) | 2 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 12 | 15
Nervous system disorders - Other, specif (Nervous system disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 5 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thromboembolic event (Vascular disorders) | 4 | 7 | 5
Injury to superior vena cava (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High TS: IROX/Bev (N=70) | High TS: FOLFOX/Bev (N=73) | Low or Indeterminate TS: FOLFOX/Bev (N=62)
Allergic reaction (Immune system disorders) | 7 | 3 | 0
Anemia (Blood and lymphatic system disorders) | 54 | 56 | 51
White blood cell decreased (Investigations) | 39 | 49 | 43
Neutrophil count decreased (Investigations) | 32 | 39 | 33
Platelet count decreased (Investigations) | 25 | 41 | 33
Hypertension (Vascular disorders) | 16 | 20 | 9
Fatigue (General disorders) | 44 | 60 | 49
Fever (General disorders) | 9 | 5 | 3
Insomnia (Psychiatric disorders) | 7 | 8 | 7
Chills (General disorders) | 5 | 7 | 6
Weight loss (Investigations) | 15 | 14 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 22 | 13
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 5 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 4 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 10 | 2
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 1 | 10 | 12
Anorexia (Metabolism and nutrition disorders) | 33 | 30 | 28
Constipation (Gastrointestinal disorders) | 20 | 23 | 21
Dehydration (Metabolism and nutrition disorders) | 7 | 8 | 6
Diarrhea (Gastrointestinal disorders) | 48 | 42 | 38
Dry mouth (Gastrointestinal disorders) | 7 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 9 | 4
Mucositis oral (Gastrointestinal disorders) | 14 | 25 | 22
Nausea (Gastrointestinal disorders) | 44 | 51 | 34
Dysgeusia (Nervous system disorders) | 14 | 23 | 14
Vomiting (Gastrointestinal disorders) | 34 | 18 | 11
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 4 | 0 | 2
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 23 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 | 29 | 29
Alkaline phosphatase increased (Investigations) | 7 | 9 | 8
Alanine aminotransferase increased (Investigations) | 4 | 5 | 1
Aspartate aminotransferase increased (Investigations) | 24 | 34 | 29
Blood bilirubin increased (Investigations) | 1 | 14 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Creatinine increased (Investigations) | 12 | 12 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 5 | 4
Hypokalemia (Metabolism and nutrition disorders) | 8 | 6 | 2
Proteinuria (Renal and urinary disorders) | 6 | 15 | 12
Hyponatremia (Metabolism and nutrition disorders) | 2 | 7 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4
Dizziness (Nervous system disorders) | 11 | 4 | 4
Anxiety (Psychiatric disorders) | 6 | 1 | 1
Depression (Psychiatric disorders) | 5 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 51 | 62 | 47
Abdominal pain (Gastrointestinal disorders) | 13 | 11 | 10
Headache (Nervous system disorders) | 6 | 11 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 11
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No